CLINICAL TRIAL: NCT02926404
Title: Evaluation of Patients Treated With Patient Specific Rods: UNiD Rods Register
Brief Title: UNiD Rods Register
Status: Terminated | Type: Observational
Why Stopped: Early terminated for administrative reasons
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 1501
Record Dates: First submitted 2016-06-27; First posted 2016-10-06 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Scoliosis; Spinal Curvatures; Spondylolisthesis; Degenerative Scoliosis
Keywords: Sagittal alignment; Surgical planning; Patient-specific; Adult Spinal Deformity
MeSH Terms: conditions — Spinal Curvatures; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric patients operated with Patient-specific rods: Patients with patient-specific rods (UNiD Rods) <18Years old
  Interventions: Device: UNiD Rods
- Adult patients operated with Patient-specific rods: Patients with patient-specific rods (UNiD Rods) >18Years old
  Interventions: Device: UNiD Rods

INTERVENTIONS:
Device: UNiD Rods — Spinal osteosynthesis
  Other Names: Patient Specific Rods

SUMMARY:
Retro-prospective study allowing inclusion of patients with spinal deformities treated by patient-specific rods (UNiD).

This study aims to assess performance, clinical outcomes and safety

DETAILED DESCRIPTION:
Despite decades of treatment and great diversity of instrumentation, the objective of sagittal spinal realignment in adult spinal deformity is achieved in only 38% of patients which reflects an inadequacy of the approach currently used.

Patient specific rods were created by Medicrea to address this gap and support surgeons in achieving what they planned to perform in terms of spinal correction based on preoperative X-rays analyses.

Beside to help surgeons in planning and to improve performance, the avoidance of manual bending is supposed to save time during surgery and to limit notches which should then reduce rod fractures responsible for surgical revisions.

A European register-like study has been set-up to assess radiological performance, clinical outcomes and revision rate following implantation of patient-specific rods in adult spinal deformities

ELIGIBILITY:
Inclusion Criteria:

* Patient operated with UNiD® Patient Specific rods from MEDICREA® INTERNATIONAL
* Patient affiliated to health care insurance (social security in France)
* Patient able to complete a self-administered questionnaire
* Patient able to sign a disclosure form or a non-opposition form

Exclusion Criteria:

* Patient not operated with Patient Specific rods from MEDICREA® INTERNATIONAL
* Pregnant patient
* Patient not affiliated to health care insurance (social security in France)
* Patient unable to sign a disclosure form
* Patient unable to complete a self-administered questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with spinal deformities
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Radiological performance compared to planning | 12 months
  The primary objective is to compare the planned sagittal parameters with those obtained postoperatively including but not limited to:
  * Sagittal vertical axis (SVA)
  * Lumbar Lordosis (LL)
  * Thoracic Kyphosis (TK)
  * Pelvic Tilt (PT)
  * Pelvic Incidence (PI)
  * Sacral Slope (SS)
  * Cobb Angle (CA)

SECONDARY OUTCOMES:
Postoperative spinal alignment | 3, 6, 12, 24 months
  Evaluation of the deformity correction in the sagittal and/or coronal plan. The primary objective is to compare the preoperative sagittal parameters with those obtained postoperatively including but not limited to:
  Sagittal vertical axis (SVA) Lumbar Lordosis (LL) Thoracic Kyphosis (TK) Pelvic Tilt (PT) Pelvic Incidence (PI) Sacral Slope (SS) Cobb Angle (CA)
Diasbility | 3, 6, 12, 24 months
  To assess patients' disability through the ODI questionnaire
Quality of life/ SRS-22 | 3, 6, 12, 24 months
  To assess patients' quality of life through the SRS-22 questionnaire
Patients' satisfaction | 3, 6, 12, 24 months
  Using a satisfaction questionnaire
Adverse event | 3, 6, 12, 24 months
  To quantify and describe adverse events
Revision | 3, 6, 12, 24 months
  To quantify and describe surgical revisions
Pain/VAS | 3, 6, 12, 24 months
  To assess patients' pain according to VAS : to 0 (better) to 10 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fiere, MD, Principal Investigator — Centre Orthopédique Santy
Locations (13):
- CH WAPI, Tournai, Belgium
- France (11):
  - Polyclinique, Bordeaux
  - Orthopôle, Bruges
  - CHU Estaing, Clermont-Ferrand
  - Hopital Saint Philibert, Lomme
  - Centre Orthopédique Santy, Lyon
  - Les Massues, Lyon
  - Hopital la Timone, Marseille
  - Hopitaux pediatriques - CHU Lenval, Nice
  - Hopital Trousseau, Paris
  - La pitié Salepetrière Hospital, Paris
  - Saint Etienne Hospital, Saint-Etienne
- Pr Andrzej Maciejczak, Tarnów, Poland

IPD SHARING:
Plan to Share IPD: No